CLINICAL TRIAL: NCT04300504
Title: Muscle in Obesity: Imaging, Function and microRNA
Status: Completed | Type: Observational
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: University of Sheffield (Other); University of Liverpool (Other)
Responsible Party: Sponsor
Other Study IDs: STH21022
Record Dates: First submitted 2019-12-19; First posted 2020-03-09 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Muscle Function
Keywords: obesity; sarcopenia; dynapenia; microRNA
MeSH Terms: conditions — Obesity; Sarcopenia | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- normal weight, not dynapenic: BMI 18.5 to 25kg/m2, waist circumference <= 88cm, healthy women aged 60-80 years, time to complete 5 chair stands <15 seconds
  Interventions: Other: observational study
- normal weight, dynapenic: BMI 18.5 to 25kg/m2, waist circumference <= 88cm,healthy women aged 60-80 years, time to complete 5 chair stands >15 seconds
  Interventions: Other: observational study
- obese, not dynapenic: BMI 30 to 40kg/m2, waist circumference > 88cm, healthy women aged 60-80 years, time to complete 5 chair stands <15 seconds
  Interventions: Other: observational study
- obese, dynapenic: BMI 30 to 40kg/m2, waist circumference > 88cm, women aged 60-80 years, time to complete 5 chair stands >15 seconds
  Interventions: Other: observational study

INTERVENTIONS:
Other: observational study — observational study

SUMMARY:
Growing evidence suggests that dynapenic abdominal obesity is associated with a greater risk of falls, functional disability and hospitalisation compared to those with dynapenia, obesity or neither phenotype. Understanding the pathogenesis underlying this phenotype has the potential to inform potential treatment strategies.

MicroRNAs can act as messengers at the cellular level to promote or block processes for muscle growth and repair, amongst other things. There is evidence that ageing changes microRNA levels in the muscle and that these changes may result in reduced muscle quality and quantity. However, it is not known whether being obese can change microRNA levels in muscle and how this relates to physical performance.

The aim of this study is to investigate the effect of dynapenic abdominal obesity on microRNA levels in serum and muscle quality and quantity in the legs of older women.

This is an observational, cross-sectional study. The investigators will recruit 4 groups of older women: normal weight, normal weight with dynapenia, obese and obese with dynapenia. The investigators will measure the microRNA levels in serum. The investigators will measure the quantity and fat content of muscle in the legs using magnetic resonance imaging. Muscle strength, fatigue and balance will be measured using gait (walking) analysis, balance tests, and a machine designed to measure leg strength and fatigue.

The investigators will measure and compare microRNA levels between groups. The investigators will use databases and computer programmes to look at all of the microRNAs which are different between groups and see how they affect the muscle. The investigators will compare muscle strength, size and fatigue between groups. The investigators will explore relationships of muscle quantity and quality measures with microRNA changes in the muscle. This approach will allow the investigators to understand how obesity affects the microRNA profile of muscle and whether this translates into impairment of function and mobility.

ELIGIBILITY:
Inclusion criteria:

* Caucasian
* Female
* BMI 18.5-25 or 30-40kg/m2
* Ages 60-80 years
* Sufficiently mobile to undergo scanning and biomechanical testing
* Able to remain motionless during scans
* Able and willing to participate in the study and provide written informed consent

Exclusion Criteria:

* BMI 18.5-25kg/m2 AND waist circumference >88cm i.e. normal weight AND abdominally obese
* BMI 30-40kg/m2 AND waist circumference <88cm i.e. obese AND not abdominally obese
* History of any long-term immobilisation (duration greater than 2 weeks in the past 12 months)
* History of hospital admission in the past 3 months
* History of recent significant weight loss (5% in 3 months or 10% in 6 months)
* Diabetes mellitus
* History of current conditions which may affect muscle metabolism

  * Malabsorption syndromes e.g. inflammatory bowel disease, pancreatic insufficiency etc.
  * Chronic renal disease
  * Diagnosed eating disorder
* Conditions which prevent the undertaking or analysis of the MRI and DXA scans or the interpretation of their results e.g. hip prosthesis, metal implants etc.
* Conditions which prevent the undertaking of the fatigue protocols e.g. hypertension etc.
* Use of medications or treatment known to affect muscle metabolism

  o Anabolic steroids, glucocorticoids, antiretrovirals etc.
* Excessive alcohol intake defined as greater than 21 units per week
* Competitive athlete, defined as participating in competitive sport at amateur or professional level
* Conditions which prevent the undertaking of a 6-minute walking test e.g. unstable angina or myocardial infarction during the previous month.

Ages: 60 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Caucasian Women Recruited from around South Yorkshire and Merseyside, UK
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-03-17 (Actual); Study Completion 2023-03-17 (Actual)

PRIMARY OUTCOMES:
Differential microRNA expression, expressed as fold-change and p-values, measured using real time quantitative polymerase chain reaction (RT-qPCR) between normal weight and obese groups, further stratified by dynapenia | 1 day (one measurement )
  Serum analyses

SECONDARY OUTCOMES:
mean difference in distance walked during 6 minute walk test between normal weight and obese, further stratified by dynapenia | 1 day (one measurement )
  6 Minute walk test
mean difference in muscle mass and volume measures between normal weight and obese, further stratified by dynapenia MRI | 1 day (one measurement )
  MRI (Magnetic Resonance Imaging)
mean difference in muscle mass and volume measures between normal weight and obese, further stratified by dynapenia DXA | 1 day (one measurement )
  DXA (dual energy X-ray absorptiometry)
mean difference in muscle strength between normal weight and obese, further stratified by dynapenia | 1 day (one measurement )
  Isokinetic dynamometer
mean difference in fatigue between normal weight and obese, further stratified by dynapenia | 1 day (one measurement )
  kinetic change in gait parameters from Opal accelerometers

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Walsh, Principal Investigator — University of Sheffield
Locations (1):
- University of Sheffield/Sheffield Teaching Hospitals, Sheffield, South Yorkshire, United Kingdom